CLINICAL TRIAL: NCT02840266
Title: The Accuracy of Automated Audiometry Application on Smart Phone to Screen Hearing Loss
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Pornthep Kasemsiri, Department of Otorhinolaryngology, Khon Kaen University
Other Study IDs: IN58320
Record Dates: First submitted 2016-07-19; First posted 2016-07-21 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
The purpose of study is to determine the diagnostic value of Hearing test program on smart phone for detected patients who has hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* Patient who underwent hearing test in our otologic clinic

Exclusion Criteria:

* Age below 15 year
* Patients who cannot following command

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient who underwent hearing test in our otologic clinic
Sampling Method: Non-Probability Sample
Enrollment: 555 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
The accuracy of automated audiometry application on smart phone to screen hearing loss | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Pornthep Kasemsiri, M.D., Principal Investigator — Khon Kaen University
Locations (1):
- Khon Kaen University, Khon Kaen, Changwat Khon Kaen, Thailand